CLINICAL TRIAL: NCT01788917
Title: Effects of Supplementation With Linseed Oil on Blood Lipids and Fatty Acid Profile in Plasma and Erythrocyte Lipids in Vegetarians
Brief Title: Effects of Supplementation With Linseed Oil on Blood Lipids in Vegetarians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Professor Dr. G. Jahreis, University of Jena
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H39_09
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2013-02

CONDITIONS: Inter-conversion n-3 PUFA, Vegetarians
Keywords: n-3 LC-PUFA, vegetarians, fatty acids, blood lipids
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vegetarians (Experimental): Dietary supplement: 10 mL linseed oil per day
  Interventions: Dietary Supplement: Linseed oil
- Omnivores (Placebo Comparator): Dietary supplement: 10 mL linseed oil per day
  Interventions: Dietary Supplement: Linseed oil

INTERVENTIONS:
Dietary Supplement: Linseed oil — Dietary supplement: 10 mL linseed oil per day

SUMMARY:
The study was performed to investigate the effects of a daily consumption of linseed oil on fatty acid distribution in plasma and red blood cell lipids and blood lipids in vegetarians.

DETAILED DESCRIPTION:
Recent studies suggest that the daily intake of n-3 LC-PUFA (EPA and DHA) can modulate cardiovascular risk factors and prevent lifestyle diseases.

The major dietary source of EPA and DHA is seafood (seaweeds and fatty cold water fishes), but they can also be found in lean red meat, in organ meats such as liver and brain. Vegetarians who do not eat meat or fish, have very low or negligible intakes of EPA (< 5 mg EPA/d) and DHA.

The purpose of the present study is to explore the tissue distribution and inter-conversion of ALA to n-3 LC-PUFA as consequence of linseed oil supplementation in vegetarians.

Eight vegetarians (3 m; 5 f) who do not eat meat, fish or seaweeds such as algae foods since least two years ago and two subjects (1 m; 1w) who consume the normal western style diet living in Jena (Germany) entered the study. The participants consumed 10 mL linseed oil per day for 10 weeks. The resulting daily dose of ALA was approx. 5.7 g/d.

ELIGIBILITY:
Inclusion Criteria:

* for the vegetarian sub-group : vegetarian diet pattern

Exclusion Criteria:

* high performance sport, daily alcohol intake and the in-take of dietary supplements (e.g., fish oil capsules)
* for the vegetarian sub-group, the consumption of fish and algae products (e.g. seaweeds, sushi)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
EPA concentrations in plasma lipids and red blood cell lipids | 10 weeks

SECONDARY OUTCOMES:
blood lipids | 10 weeks
  total cholesterol, triacylglycerides, high density cholesterol, low density cholesterol, lipoprotein a

OTHER OUTCOMES:
parameters of iron status | 10 weeks
  transferrin, ferritin, transferrin saturation, total ferritin